CLINICAL TRIAL: NCT02187874
Title: Timing of Umbilical Cord Occlusion in Premature Babies( <33 w). Delayed vs Early.
Acronym: CODE-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR(AMI)18/2014; PR(AMI)18/2014 (Other: Hospital Universitari Vall d'Hebron Research Institute)
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Delayed Umbilical Cord Clamping Benefits; Postpartum Haemorrhage; Intraventricular Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early umbilical cord occlusion (Active Comparator): Cord clamping will be performed before 30 seconds after delivery, annoting the exact time of clampage and initiating reanimation and postnatal care procedures as usual. 60 second after delivery of the new born, 10 IU of Oxytocin will be administered intramuscularly.
  Interventions: Procedure: early umbilical cord occlusion; Drug: Oxytocin
- delayed umbilical cord occlusion (Experimental): One of the paediatricians will hold the newborn ( in vaginal deliveries between 20-30 cm under the mother, in C-sections between the legs of the mother) until clamping of the umbilical cord is indicated by a second paediatrician who will be controlling the time and overall state of the baby. The baby will be wrapped during this time in a thermal blanket in a flexed lateral decubitus position to minimise stress and heat loss. Time of clamping: after 30 to 60 seconds( preferably 60). If loss of the baby's wellbeing is suspected, the paediatrician will assess the newborn's heart rate , stopping the procedureif this falls under 100ppm, initiating at that moment the necessary reanimation procedures.
  60 second after the delivery of the new born 10 IU of oxytocin will be administered intramuscularly.
  Interventions: Procedure: delayed umbilical cord occlusion; Drug: Oxytocin

INTERVENTIONS:
Procedure: delayed umbilical cord occlusion
  Arms: delayed umbilical cord occlusion
Procedure: early umbilical cord occlusion
  Arms: early umbilical cord occlusion
Drug: Oxytocin

SUMMARY:
Early cord clamping after delivery has been common practice for many decades as part of the active management of the third stage of labour. However in recent years, several studies have shown that delayed cord clamping may offer important benefits to the newborn. The data gathered indicate that delayed cord clamping may be particularly useful in premature babies, between 26 and 32 weeks of gestational age, reducing the need for blood transfusion and the incidence of intraventricular haemorrhage.

However it is argued that the described potential benefits of delayed cord clamping could be negated by the increased risk of polycythaemia and jaundice in the newborn, as well as by potential interference with the postpartum haemorrhage management, initial care and reanimation of the premature newborn, and the possibility of cord blood donation. These factors, together with as the lack of homogeneity among existing studies regarding the delayed cord clamping technique create the need, in our opinion, for further research, to establish the proper place of this measure.

Our hypothesis is that delayed cord clamping in the premature newborn significatively reduces the need for blood transfusions and intraventricular haemorrhage, compared with usual early cord clamping.

Secondary outcomes:

* To define the impact of delayed cord clamping on neonatal assessment parameters after delivery: APGAR score, cord pH, need for mechanical ventilation or reanimation.
* Neonatal mortality and morbidity
* Effect of the procedure on the incidence and severity of maternal postpartum haemorrhage
* To study the correlation between Iron metabolism and reticulocitary haemoglobin levels in cord and infant blood.

ELIGIBILITY:
Inclusion Criteria:

* Deliveries ( either vaginal or by C-section) between 26 and 32.6 weeks of gestation.
* Patients must be over 18 years old.
* Patient understands and signs informed consent.

Exclusion Criteria:

* Urgent C-section
* gestational age under 22 or over 33 weeks
* Major fetal anomalies (requiring surgery or with a high risk of neonatal death or incapacity)
* Major uterine malformations
* Placenta previa.
* Multiple gestations
* Fetal hydrops
* Severe Iso- Immunization
* HIV-positive mother
* Severe Intrauterine growth restriction ( Reverse atrial Flow in DV)
* Intrauterus Ventricular haemorrhage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of red blood cell transfusions to the newborn | for the duration of hospital stay, an expected average of 2 months.
Intraventricular Haemorrhage incidence | from delivery, for the duration of hospital stay, an expected average of 2 months.
Maternal postpartum haemorrhage incidence | within 24 hours after birth
Volume of neonatal red blood cell transfusions | for the duration of hospital stay, an expected average of 2 months.

SECONDARY OUTCOMES:
Neonatal mortality | up to 27 days after birth.
  * early ( 0 to 6 days after birth)
  * late ( 7 to 27 days after birth)

OTHER OUTCOMES:
APGAR score | 10 minutes after delivery
Umbilical cord blood pH | 0-15 minutes after delivery
Neonatal intubation | 0-30 minutes after delivery
Incidence of intensive reanimation of the newborn | 0-30 minutes after delivery
  Use of vasoactive drugs.
Incidence of adverse events during hospital stay of the newborn. | for the duration of hospital stay, an expected average of 2 month.

CONTACTS AND LOCATIONS:
Overall Officials: Melchor Carbonell Socias, MD, Principal Investigator — Hospital Vall d'Hebron; Angela Gregoraci, MD, Principal Investigator — Hospital Vall d'Hebron; Maria Goya Canino, MD, Study Director — Hospital Vall d'Hebron; Maria Angeles Linde, MD, Study Director — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari de la Vall d'Hebron, Barcelona, Barcelona, Spain